CLINICAL TRIAL: NCT05007704
Title: Competencies Required by Anesthesiologists Managing Critically Ill Medical and Surgical Patients in an Intensive Care Unit
Brief Title: Competencies Required by Anesthesiologists Managing Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Prashant Nasa (Other)
Collaborators: World Federation of Societies of Anaesthesiologists (Unknown)
Responsible Party: Sponsor-Investigator, Prashant Nasa, Head Critical Care Medicine, NMC Specialty Hospital
Organization: NMC Specialty Hospital (Other)
Other Study IDs: WFSA-CCM
Record Dates: First submitted 2021-08-11; First posted 2021-08-16 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Training; Education; Competence
Keywords: Training of Anesthesiologists; Training in Intensive care medicine; Anesthesiologists intensivist; Curriculum of training for Anesthesiologists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anesthesiologists for preliminary survey: Anesthesiologists who have completed their training within the last three years to identify preliminary competencies for Delphi round one survey.
- Global Experts in Anesthesiology and Critical Care Medicine: Anesthesiologist (a medical graduate who has completed a nationally recognized Anesthesiology training programme) involved in the management of critically ill patients in ICU and have more than ten years of experience in teaching and training in Critical Care. They will be involved in the Delphi process to generate expert consensus on the additional competencies (mandatory desirable and optional) required for Anesthesiologists to practice Critical Care in the Intensive Care Unit (ICU).
  Interventions: Behavioral: Global Experts Consensus opinion using Delphi Methodology

INTERVENTIONS:
Behavioral: Global Experts Consensus opinion using Delphi Methodology — The Investigators will conduct iterative Delphi Rounds with Global experts to achieve consensus on Competencies required for Anesthesiologists to manage critically ill medical and surgical patients in ICU
  Groups: Global Experts in Anesthesiology and Critical Care Medicine

SUMMARY:
Critical Care Medicine (CCM) has emerged as an independent specialty over the last few decades. Anesthesiologists being perioperative physicians, often practice CCM full time or part-time. Deficiencies have been noted by experts in the Anesthesiology training in certain competencies required for the management of critically ill medical and surgical patients in the Intensive care unit (ICU). This is often compounded by considerable variation in the training curriculum of the Anesthesiologists based on the geographical region and base specialty. The Intensive & Critical Care Medicine Committee of the World Federation of Societies of Anesthesiologists (WFSA), has developed a preliminary survey of recently qualified Anesthesiologists, to review the existing competencies for CCM in the Anesthesiology curriculum across the globe. The results of this survey will be used to identify the gaps and additional competencies required for Anesthesiologists to practice Critical Care in ICU through expert consensus, using a Delphi process.

DETAILED DESCRIPTION:
BACKGROUND:

CCM has emerged as an independent specialty over the last few decades. Anesthesiologists being perioperative physicians are an integral part of this progress, with many of them opting for CCM as a full-time career. The coronavirus disease 2019 (COVID-19) pandemic has brought unprecedented challenges to the health care system. Anesthesiologists working in the operating room (OR) and those working in the ICU have been the frontline workers along with other Critical Care professionals in the management of critically ill patients with COVID-19. Though a few countries have recognized CCM as a separate specialty of medicine, in most countries, it is considered as a sub-specialty of broad specialties like Anesthesiology, Pulmonary Medicine or Internal Medicine. Some professional bodies have developed a formal curriculum for training in CCM. The Competency-Based Training programme in Intensive Care Medicine (CoBaTrICE) from the European Society of Intensive Care Medicine (ESICM) is a widely accepted formal structured training curriculum in CCM. Most curricula are designed only for high-income, well-resourced training and practice environments and do not account for additional skills and competencies that may be required to practice in resource variable settings, something the COVID-19 pandemic has demonstrated needs to be universal. The transition of Anesthesiologists working in OR or managing critically ill surgical/ polytrauma patients into working in ICU has largely been smooth. Nevertheless, experts have noted deficiencies in the Anesthesiology training in certain competencies required for the management of critically ill medical and surgical patients in the ICU. This is often compounded by considerable variation in the training curriculum of the Anesthesiologists based on the geographical region and type of institution. There is a need to identify these competencies so that Anesthesiologists who wish to practice full time or part-time Critical Care can acquire these competencies to improve their ability to manage critically ill patients in ICU in different World Health Organization defined healthcare facilities levels. This may also help provide guidance to educators worldwide regarding the competencies to be included in Anesthesiology training that may help Anesthesiologists work better with critically ill patients in ICU. These competencies have never been formally identified or published. The investigators plan to review the existing competencies for CCM in the Anesthesiology curriculum across the globe through a preliminary survey. Thereafter, the investigators plan to identify the additional competencies required through consensus among Experts, using a Delphi method. These additional competencies, classified as mandatory, desirable, and optional, may serve as a guide for Anesthesiologists to practice Critical Care in ICU in different levels of health care facilities worldwide.

OBJECTIVES

1. The investigators aim to review/identify the existing competencies for CCM in the Anesthesiology curriculum across the globe.
2. The investigators aim to generate expert consensus on the additional competencies (mandatory desirable and optional) required for Anesthesiologists to practice Critical Care in the ICU.
3. Provide guidance to educators worldwide regarding the competencies to be included in the Anesthesiology curriculum that may help Anesthesiologists work better with critically ill patients in ICU.

METHODOLOGY

Steering Committee:

A Steering Committee comprising of Anesthesiologists with experience in CCM will be formed under the auspices of the Intensive and Critical Care Medicine Committee (ICCCM) of the World Federation of Societies of Anaesthesiologists (WFSA).

Preliminary survey:

The Steering Committee will develop a preliminary survey to assess the knowledge and skills of Anesthesiologists across the globe following Anesthesiology training, which is required to achieve the various Critical Care competencies. A literature review on the existing Critical Care competencies from various professional bodies will be conducted to develop a list of Critical Care competencies, using CoBaTrICE as a base. The preliminary survey will be sent to approximately 500 Anesthesiologists across the globe by the Experts. The competencies of participants in CCM will be assessed under six domains in the survey (Disease diagnosis and management, Procedures, Monitoring and therapeutic interventions, Resuscitation, Communication and End-of-life care, Patient safety and Crisis Resource Management) using a 5-point Likert scale (never seen, have observed, can manage under supervision, can manage with minimal assistance, and can manage independently).

The first section of this survey will include the participant demographics, country of origin and training, year of completing training, and a few training characteristics. The results of the survey will be used to draft competencies for inclusion in Round one of the Delphi.

Delphi process:

The Delphi process is a well-established methodology to generate consensus on a particular topic using the "collective intelligence" of panel members. The steering committee members will perform a literature search on the available evidence, draft the initial statements and conduct iterative Delphi rounds to generate consensus among the experts. The Steering Committee members will not participate in the Delphi surveys themselves.

Steps of the Delphi process

Step 1: Establishing a preliminary list of competencies:

A literature review on the existing Critical Care competencies from various professional bodies will be conducted to develop a list of Critical Care competencies, using CoBaTrICE as a base and categorized under the six core domains (disease diagnosis and management, procedures, monitoring and therapeutic interventions, resuscitation, communication and end-of-life care, patient safety and crisis resource management). The results of the preliminary survey will be used to draft statements for Round one of Delphi.

Step 2: Preparation of the Delphi Round one survey:

The list of the competencies will be sent to the Experts as a Delphi questionnaire. The anonymity of the participating experts will be maintained during the Delphi rounds. The participant will be asked to score each of the competencies listed on a 5-point Likert scale (non-essential, optional, optional but desirable, desirable, and mandatory). The participating expert will be invited to provide feedback regarding omission, addition, or modification of the items on the questionnaire. The response and feedback of experts will be collated during the analysis of results and shared in the following survey as controlled feedback.

Step 3: Subsequent Delphi Rounds:

The steering committee will review the results of round one. The competencies listed will be modified, deleted, or added if found ambiguous based on the feedback and comments of the results. Competencies deemed "non-essential" by more than 50% of the respondents will be eliminated. The remaining competencies will be continued in the subsequent rounds until consensus is achieved (>80% of respondents). Lower-rated items identified for removal may be retained in the second round if more than 20% of participating experts considered them "mandatory". The summary results of Round two will be presented to Experts, and the survey process will be repeated with the modified questionnaire. The Delphi rounds will be continued till desired consensus and stability is achieved for competencies.

Step 4: Final Consensus on Competencies to be included:

The summary results of the last stable round will be used to issue the consensus on the additional competencies to be included. These competencies will also be classified as those mandatory, desirable, and optional, which may serve as a guide to decide which competencies are required for working in different levels of health care facilities worldwide. The results of the final survey, consensus competencies, and the manuscript will be circulated among the experts for approval before submission for publication.

ELIGIBILITY:
Inclusion Criteria:

Preliminary survey

• Anesthesiologists who have completed their training within the last three years.

Selection of experts for the Delphi process:

* Anesthesiologist (a medical graduate who has completed a nationally recognized Anesthesiology training programme)
* Involved in the management of critically ill patients in ICU
* More than ten years of experience in teaching and training in Critical Care.

Exclusion Criteria:

Preliminary survey

* Anesthesiologists have started training in critical care medicine immediately after completion of their Anesthesia training
* Anesthesiologists who refused to participate

Delphi Process selection of experts:

* Non-Anesthesiologist intensivist
* Anesthesiologist not involved in the management of critically ill patient
* Pediatric Intensivist

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Preliminary survey: A cross-sectional will be circulated through snowball sampling technique among Anesthesiologists worldwide.
  Delphi Process:
  Global Experts in Anesthesiology and Critical Care Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 1155 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Development of Preliminary Competencies | 30 days
  Using a 5-point likert scale (never seen, have observed, can manage under supervision, can manage with minimal assistance, and can manage independently) through a cross-sectional survey with 500 recently (less than three years) trained Anesthesiologists.
Consensus among participating experts | 45 days
  The participating experts will be asked to score each of the competencies listed on a 5-point Likert scale (nonessential, optional, optional but desirable, desirable, and mandatory).The Delphi rounds will be continued till desired consensus and stability is achieved for competencies.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila N Myatra, MD, Principal Investigator — Tata Memorial Hospital, Mumbai, India
Locations (1):
- Tata Memorial Hospital, Mumbai, India

IPD SHARING:
Plan to Share IPD: Undecided
The study protocol and statistical analysis of preliminary survey and Delphi process

REFERENCES:
- [Background] Hastie J. Anesthesiologists as perioperative leaders. Int Anesthesiol Clin. 2020 Fall;58(4):58-63. doi: 10.1097/AIA.0000000000000296. No abstract available. PMID 32889956
- [Background] Barrett H, Bion JF. An international survey of training in adult intensive care medicine. Intensive Care Med. 2005 Apr;31(4):553-61. doi: 10.1007/s00134-005-2583-7. Epub 2005 Mar 5. PMID 15750798
- [Background] CoBaTrICE Collaboration. The educational environment for training in intensive care medicine: structures, processes, outcomes and challenges in the European region. Intensive Care Med. 2009 Sep;35(9):1575-83. doi: 10.1007/s00134-009-1514-4. Epub 2009 Jun 23. PMID 19547957
- [Background] Kain ZN, Fitch JC, Kirsch JR, Mets B, Pearl RG. Future of anesthesiology is perioperative medicine: a call for action. Anesthesiology. 2015 Jun;122(6):1192-5. doi: 10.1097/ALN.0000000000000680. No abstract available. PMID 25886775
- [Background] Gelb AW, Morriss WW, Johnson W, Merry AF, Abayadeera A, Belii N, Brull SJ, Chibana A, Evans F, Goddia C, Haylock-Loor C, Khan F, Leal S, Lin N, Merchant R, Newton MW, Rowles JS, Sanusi A, Wilson I, Velazquez Berumen A; International Standards for a Safe Practice of Anesthesia Workgroup. World Health Organization-World Federation of Societies of Anaesthesiologists (WHO-WFSA) International Standards for a Safe Practice of Anesthesia. Anesth Analg. 2018 Jun;126(6):2047-2055. doi: 10.1213/ANE.0000000000002927. PMID 29734240
- [Background] Diamond IR, Grant RC, Feldman BM, Pencharz PB, Ling SC, Moore AM, Wales PW. Defining consensus: a systematic review recommends methodologic criteria for reporting of Delphi studies. J Clin Epidemiol. 2014 Apr;67(4):401-9. doi: 10.1016/j.jclinepi.2013.12.002. PMID 24581294
- [Background] Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to decide its appropriateness. World J Methodol. 2021 Jul 20;11(4):116-129. doi: 10.5662/wjm.v11.i4.116. eCollection 2021 Jul 20. PMID 34322364
- [Background] Junger S, Payne SA, Brine J, Radbruch L, Brearley SG. Guidance on Conducting and REporting DElphi Studies (CREDES) in palliative care: Recommendations based on a methodological systematic review. Palliat Med. 2017 Sep;31(8):684-706. doi: 10.1177/0269216317690685. Epub 2017 Feb 13. PMID 28190381

DOCUMENTS (1):
  • Study Protocol (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT05007704/Prot_000.pdf